CLINICAL TRIAL: NCT06444321
Title: INTEgRated Health CARE for Patients With Frailty and Heart Failure (INTERCARE-HF): Evaluation of an Innovation Project
Brief Title: INTEgRated Health CARE for Patients With Frailty and Heart Failure
Acronym: INTERCARE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Drammen municipality (Unknown); University of Oslo (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 678261
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure; Frailty; Frail Elderly Syndrome; Symptom, Behavioral; Utilization, Health Care; Quality of Life
MeSH Terms: conditions — Heart Failure; Frailty; Behavioral Symptoms; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Open intervention study with a matched control-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A structured, person-centred and coordinated treatment and follow-up plan tailored to co-morbidities, risk areas, cognitive function and functional level, and the patients' symptoms and needs will be developed by an interdisciplinary team from the hospital and the primary care service. The closest relatives were encouraged to participate. The plan will be followed-up and evetually adjusted after one week and then at least monthly by nurses in the municipality through phone calls and /or home visits. A detailed description will be manualized in a handbook.
  Interventions: Behavioral: INTERCARE-HF
- Matche control group (Active Comparator): A matched control-group will be recruited from the ongoing IT-HEART RCT
  Interventions: Behavioral: INTERCARE-HF

INTERVENTIONS:
Behavioral: INTERCARE-HF — Develpent of an individualized treatment and follow-up plan tailored to co-morbidities, risk areas, cognitive function and functional level as well as the patients' symptoms and needs.
  Other Names: Matched control group

SUMMARY:
Frailty, an aging-related syndrome of physiological decline characterized by marked vulnerability to adverse health outcomes, has attracted increasing attention in cardiology due to the growing elderly population with heart failure. Frail patients are mainly excluded from large cardiovascular intervention studies, and clinical trials addressing frailty and showing an impact on treatment on symptom burden, quality of life and /or outcome has been requested in recent guidelines and consensus documents. The INTEgrRated health CARE for patients with severe frailty and Heart Failure (INTERCARE-HF) is a proof-of-concept study that aims to evaluate the effect of integrated healthcare services for heart failure patients with a severe level of frailty by establishing interdisciplinary and coordinated follow-up teams across the healthcare boundaries. These teams will assess the patient's needs, goals, and risk areas, conduct advance care planning, and develop individualized treatment and follow-up plans. An open-label, non-randomized intervention study aims to recruit 20 patients and heart failure and a clinical Frailty Score (CSF) >=5. A control-group (N=40) matched on age an clinical frailty scale score will be included. The overall hypothesis is that the intervention is feasible in routine clinical practice with favorable effects on quality of life, symptoms, caregiver distress, and healthcare service utilization.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Admitted to hospital with heart failure with symptoms of decompensation including dyspnoea in NYHA class ≥ II, pulmonary congestion on chest x-ray and/or other signs like oedema or positive rales on auscultation and elevated NT-proBNP concentrations at screening
* Clinical Frailty Score ≥5
* Signed informed consent by patient and closest relatives* and expected cooperation according to the protocol, ICH/GCP and national/local regulations

  * Although we preferably will recruit both patients and their relatives, participation from the next-of-kin will not be an exclusion criterium.

Exclusion Criteria:

* Inability to comply with all study requirements, due to major co-morbidities or psychosocial issues, or a history of noncompliance, that might compromise the patient's ability to understand and/or comply with the protocol instructions or follow-up procedures.
* Not being able to understand Norwegian.
* Permanent nursing home and estimated to stay alive for less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in symptom control and patient satisfaction | From baseline to weeks 6, 12, and 52
  Between-group differences in The Edmonton Symptom Assessment System revised (ESAS-r) scores
Changes in health-related quality of life | From baseline to weeks 6, 12, and 52
  Between-group differences in Kansas City Cardiomyopathy Questionnaire 12 scores

SECONDARY OUTCOMES:
Changes in caregiver distress | From baseline to weeks 6, 12, and 52
  Changes in Relatives Stress Scale (RSS) scores
Total number of days lost due to unplanned hospital re-admissions during the follow-up | From baseline to weeks 6, 12, and 52
  Differences in the percentage of days out of the total number of days lost due to unplanned hospital admissions
The number of days lost due to unplanned hospital re-admissions for specific diagnosis during the follow-up | From baseline to weeks 6, 12, and 52
  Differences in the percentage of days out of the number of days lost due to unplanned hospital admissions for i. heart failure, ii. kidney failure, dehydration or hyper/hypokalemia, iii. Falls and fractures
Total number of hospitalizations | From baseline to weeks 6, 12, and 52
  Differences in the total number of hospitalizations during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Drammen Hospital, Drammen, Akershus, Norway